CLINICAL TRIAL: NCT07258277
Title: Comparative Study Between Adductor Canal Block With IPACK (Infiltration Between the Popliteal Artery and Capsule of the Knee) Versus Genicular Nerves Block With IPACK for Post-operative Analgesia in Knee Arthroscopy
Brief Title: Adductor Canal Block With IPACK Versus Genicular Nerves Block With IPACK for Post-operative Analgesia
Acronym: IPACK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Gehad Fathy Mohamed Sadek, Lecturer of Anesthesiology and ICU, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1391
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Postoperative Analgesia
Keywords: IPACKL/ adductor canal block/ genicular nerves block
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Intervention Model Description: This prospective randomized controlled clinical study will be conducted in anesthesiology and intensive care department at Minia University Hospital (MUH) on 72 adult patients of both genders, aged between 20 years to 70 years old, ǀ and ǀǀ classification of The American Society of Anesthesiologists (ASA) planned to undergo elective unilateral knee surgeries under spinal anesthesia.Our 72 patients were randomly divided into 3 groups, each group includes 24 patients
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IA (IPACK with adductor cannal block) (Active Comparator): receive ultrasound-guided IPACK block in supine position with externally rotated leg and flexed knee, 15 ml of 0.25% plain bupivacaine then another 15 ml of 0.25% plain bupivacaine at the mid-thigh for the ACB.
  Interventions: Other: IPACK with adductor canal block
- IG (IPACK with genicular nerves block) (Active Comparator): receive ultrasound-guided IPACK block in supine position with externally rotated leg and flexed knee, 15 ml of 0.25% plain bupivacaine then at the anterior surface of the knee 16 ml of 0.25% plain bupivacaine divided on the 4 genicular nerves (superior medial, superior lateral, inferior medial and inferior lateral).
  Interventions: Other: IPACK with Genicular nerves block
- C (Spinal block) (Active Comparator): won't receive any nerve block, only spinal anesthesia.
  - Then spinal anesthesia will be given to all patients in the three groups, 3 ml (15 mg) 0.5% hyperbaric bupivacaine will be administered intrathecal at level of L3-4 or L4-5 interspace.
  Interventions: Other: Spinal Block

INTERVENTIONS:
Other: IPACK with adductor canal block — receive ultrasound-guided IPACK block in supine position with externally rotated leg and flexed knee, 15 ml of 0.25% plain bupivacaine then another 15 ml of 0.25% plain bupivacaine at the mid-thigh for the ACB.
  Arms: IA (IPACK with adductor cannal block)
Other: IPACK with Genicular nerves block — receive ultrasound-guided IPACK block in supine position with externally rotated leg and flexed knee, 15 ml of 0.25% plain bupivacaine then at the anterior surface of the knee 16 ml of 0.25% plain bupivacaine divided on the 4 genicular nerves (superior medial, superior lateral, inferior medial and inferior lateral).
  Arms: IG (IPACK with genicular nerves block)
Other: Spinal Block — won't receive any nerve block, only spinal anesthesia.
  - Then spinal anesthesia will be given to all patients in the three groups, 3 ml (15 mg) 0.5% hyperbaric bupivacaine will be administered intrathecal at level of L3-4 or L4-5 interspace.
  Arms: C (Spinal block)

SUMMARY:
In our study, we will find out the efficacy of those peripheral nerve blocks on postoperative pain in knee arthroscopy.

The aim is to evaluate the efficacy of combined ultrasound-guided IPACK with adductor canal nerve block versus ultrasound-guided IPACK with genicular nerves block on postoperative pain in knee arthroscopy.

DETAILED DESCRIPTION:
Effective perioperative pain treatment has been documented to facilitate accelerated rehabilitation and recuperation, hence providing improved functional outcomes among individuals following knee surgeries. As a result, there has been a need to create multimodal analgesic regimens that include the usage of both regional anesthetic and systemic analgesics (Society, 2012).

Management of pain for knee surgery has been challenging, where various methods like epidural, peripheral nerve block (PNB), Local Infiltration Analgesia (LIA), intravenous (IV) analgesics like opioids, non-steroidal anti-inflammatory drugs (NSAIDs) and intra-articular (IA) injections, have been used (Tian et al., 2020).

In knee surgeries, the most difficult factor to control is pain, but early movement following surgery can be facilitated by motor-sparing regional anesthetic blocks and ultrasound-guided nerve blocks (Leung et al., 2018).

Perioperative multimodal analgesic strategies, consisting of "motor-sparing" regional anesthetic techniques combined with systemic nonopioid medications that target various pain pathways, have been developed to mitigate this risk; they confer improved pain scores and patient satisfaction, reduced opioid consumption and opiate-related adverse effects, early postoperative ambulation, shortened hospital stay, and fewer surgical complications (Kandarian et al., 2019).

The adductor canal block (ACB) is a regional anesthesia technique used to provide analgesia to the anterior and medial areas of the thigh and the knee (El-Boghdadly et al., 2021).

The ACB targets the nerves that pass through the adductor canal. The primary nerve target of the ACB is the saphenous nerve, a branch of the femoral nerve. The saphenous nerve is responsible for the sensitive innervation of the leg's medial section, from the knee to the ankle. In addition to the saphenous nerve, the ACB may also block the anterior branches of the obturator nerve and the medial femoral cutaneous nerve, which supply sensation to the medial section of the thigh (Woodworth et al.,2023).

Often, it is challenging to adequately anesthetize the posterior knee through regional technique for postoperative analgesia. Local anesthetic infiltration of the interspace between the popliteal artery and capsule of the posterior knee, known as the IPACK block, can be used to reduce pain after knee surgery. The IPACK block is a novel regional technique developed to provide analgesia to this area without compromising motor function (Elliott & Thobhani, 2014).

The IPACK, combined with ACB, involves blocking the sensory nerves of the anterior, medial, and posterior knee, preserving motor function to encourage early ambulation and expedited rehabilitation (Sankineani et al., 2018).

The genicular nerves include branches from the femoral, common peroneal, saphenous, tibial, and obturator nerves which innervate the knee capsule (Kim et al., 2018).

The superolateral, superomedial, and inferomedial branches of the genicular nerve were reported to be in proximity to the periosteum of tibia and femur, and the superolateral, inferolateral, superomedial, and inferomedial quadrants of the anterior knee joint were shown to be innervated by superior lateral, inferior lateral, superior medial and inferior medial branches of the genicular nerve, respectively alongside the branches of peroneal and femoral nerves (Tran et al., 2018).

A genicular nerve block specifically targets these branches for postoperative analgesia in knee surgery.

First analgesic request (to evaluate the efficacy of combined ultrasound-guided IPACK with adductor canal nerve block versus ultrasound-guided IPACK with genicular nerves block on postoperative pain in knee arthroscopy) is the primary outcome of the study.

VAS score (dynamic and static), Hemodynamics (heart rate, blood pressure and SpO2), Total analgesic requirements, Time Up and Go test (for calculating time of postoperative movement) and Complications as (Nausea, vomiting, Allergy, Tachycardia, Hypotension or Local anesthetic toxicity) are the secondery outcomes.

Neurological deficiencies prior to surgery, Severe Cardiovascular, renal, hepatic comorbidities, Hematological disorders, abnormal coagulation parameters, Psychiatric illnesses, opioid addiction or Allergies to any of the medications will be utilized in the study will be excluded.

A prospective randomized controlled clinical study will be conducted in anesthesiology and intensive care department at Minia University Hospital (MUH) on 72 adult patients of both genders, aged between 20 years to 70 years old, ǀ and ǀǀ classification of The American Society of Anesthesiologists (ASA) planned to undergo elective unilateral knee surgeries under spinal anesthesia.

Patients will be divided into 3 groups, each group includes 24 patients:

ELIGIBILITY:
Inclusion Criteria:

* ASA l & ll
* planned to undergo elective unilateral knee surgeries under spinal anesthesia
* age between 20 to 70 years old
* both sex

Exclusion Criteria:

* Patient refusal
* Neurological deficiencies prior to surgery
* Severe Cardiovascular, renal and hepatic comorbidities
* Hematological disorders and abnormal coagulation parameters
* Psychiatric illnesses and opioid addiction
* Allergies to any of the medications will be utilized in the study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
first analgesic request | within 24 hours
  the first time the patient will ask analgesia postoperative

SECONDARY OUTCOMES:
Changes in Visual Analogue Score | To be measured immediately postoperative, 2h later, 4h, 6h, 8h, 12h, 18h, 24h
  measuring pain intensity on a ruler with a score ranging from 0-100 mm (Weigl & Forstner, 2021).
  * Dynamic: during the movement of the patient
  * Static: while the patient is bed ridden.
    * No pain: 0-4 mm
    * Mild pain: 5-44 mm
    * Moderate pain: 45-74 mm
    * Severe pain: 75-100 mm,
Total analgesic requirement | within 24 hours
  dose of fentanyl or paracetamol will be used postoperative
Time Up and Go Test (TUG) | postoperative: 6h, 12h, 18h and 24h.
  * Ask the patient to get up from a chair
  * Then walk three meters, turn and return back to the chair
  * Finally, sit on the chair again
  * We calculate the time spent during the movements of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Gehad Fathy Sadek, MD, Principal Investigator — Minia University
Locations (1):
- Minia University Hospital, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No